CLINICAL TRIAL: NCT01885845
Title: A Comparison of the Excellent BRASSS-V Drape™ and an Indirect Blood Measurement Protocol for the Measurement of Blood Loss During Third Stage of Vaginal Delivery
Brief Title: Excellent BRASSS-V Drape™ Versus Indirect Measurement Protocol for Measurement of Postpartum Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2.4.7
Record Dates: First submitted 2013-06-19; First posted 2013-06-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum blood loss measurement; BRASSS-V drape
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BRASSS-V drape (Experimental): Immediately after delivery and cord clamping, blood measurement will begin. The calibrated delivery drape should be placed under the buttocks of the woman and tied around the woman's waist with the funnel portion hanging down between her legs. Blood loss will be measured for at least one hour or, if bleeding continues after one hour, until active bleeding has stopped.
  Interventions: Device: Excellent BRASSS-V Drape™.
- Indirect weight method (Experimental): Just after delivery and cord clamping, a sheet with plastic backing will be placed under the buttocks of the woman. A basin will be placed directly under her on a small shelf on the delivery table. Blood loss will be measured for at least one hour or, if bleeding continues after one hour, until active bleeding has stopped.
  After bleeding has stopped, all gauze pieces and mops will be counted and then placed in the collection basin. The basin will be placed on the scale and weighed. The weight of the blood will be assessed by subtracting the weight of the basin, gauzes and mops from the total weight of the soaked materials assuming that one gram is equivalent to 1 ml.
  Interventions: Other: Indirect weight assesment of blood loss

INTERVENTIONS:
Device: Excellent BRASSS-V Drape™. — Immediately after delivery and cord clamping, blood measurement will begin. The calibrated delivery drape should be placed under the buttocks of the woman and tied around the woman's waist with the funnel portion hanging down between her legs. Blood loss will be measured for at least one hour or, if bleeding continues after one hour, until active bleeding has stopped.
  Arms: BRASSS-V drape
Other: Indirect weight assesment of blood loss — Just after delivery and cord clamping, a sheet with plastic backing will be placed under the buttocks of the woman. A basin will be placed directly under her on a small shelf on the delivery table. Blood loss will be measured for at least one hour or, if bleeding continues after one hour, until active bleeding has stopped.
  After bleeding has stopped, all gauze pieces and mops will be counted and then placed in the collection basin. The basin will be placed on the scale and weighed. The weight of the blood will be assessed by subtracting the weight of the basin, gauzes and mops from the total weight of the soaked materials assuming that one gram is equivalent to 1 ml.
  Arms: Indirect weight method

SUMMARY:
Postpartum hemorrhage is one of the most common causes of maternal mortality and serious maternal morbidity, especially in the developing world. In India, hemorrhage is a major cause of maternal mortality: A study by the Register General in 1993 showed that 23 percent of all maternal deaths in rural areas were caused by hemorrhage (Sibley, 2005).

The measurement of postpartum blood loss and identification of postpartum hemorrhage are important measures in efforts to prevent and treat postpartum hemorrhage. In recent years, researchers have employed several different methods to measure blood loss in hospital and community-based birth settings. Although research has demonstrated that these laboratory measures are more accurate then visual estimation techniques, no studies have explicitly documented the systematic differences (if any) among different collection modalities. Moreover, only a few of these studies have correlated measured blood loss with changes in hemoglobin levels experienced between the antepartum and postpartum period. The aim of this study is to compare variations in the measurement of blood loss obtained using two popular measurement methods: the Excellent BRASSS-V Drape™ and a modified version of the blood collection method developed by the World Health Organization (WHO).

DETAILED DESCRIPTION:
Postpartum hemorrhage is one of the most common causes of maternal mortality and serious maternal morbidity, especially in the developing world. In India, hemorrhage is a major cause of maternal mortality: A study by the Register General in 1993 showed that 23 percent of all maternal deaths in rural areas were caused by hemorrhage (Sibley, 2005).

The measurement of postpartum blood loss and identification of postpartum hemorrhage are important measures in efforts to prevent and treat postpartum hemorrhage. However, visual estimation of postpartum hemorrhage often leads to underestimation of blood loss and subsequent delays in the seeking or provision of appropriate treatment. In recent years, researchers have employed several different methods to measure blood loss in hospital and community-based birth settings. Although research has demonstrated that these laboratory measures are more accurate then visual estimation techniques, no studies have explicitly documented the systematic differences (if any) among different collection modalities. Moreover, only a few of these studies have correlated measured blood loss with changes in hemoglobin levels experienced between the antepartum and postpartum period. The aim of this study is to compare variations in the measurement of blood loss obtained using two popular measurement methods: the Excellent BRASSS-V Drape™ and a modified version of the blood collection method developed by the World Health Organization (WHO).

We propose a randomized prospective study to compare the measurement of blood loss during the third stage of labor with two different methods: the modified WHO blood measurement protocol and the Excellent BRASSS-V Drape™. Upon admission in the labor ward, study staff will approach all delivering women about participation in the study and seek informed consent. Blood loss will be measured for all consenting women with vaginal deliveries.

Women who agree to participate will be randomized to one of two blood collection techniques: a modified version of the WHO blood measurement protocol or the Excellent BRASSS-V Drape™. Blood loss will be measured from immediately after delivery and cord clamping for a period of at least one hour or until active bleeding stops. The blood loss will then be quantified by the study staff and recorded on the study form. Women will receive the facility's standard care for the management of the third stage of labor and, if applicable, treatment of PPH.

Measures of postpartum hemoglobin levels will be taken at admission for delivery and twenty-four hours post-delivery for a randomly selected sub-set of study participants. Besides the measurement of blood loss and the regular measurement of hemoglobin for a sub-sample of participants, there will be no change to the hospital's standard procedures for labor and delivery.

ELIGIBILITY:
Inclusion Criteria:

• Vaginal birth

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Mean blood loss | after delivery to when active bleeding has stopped or at least one hour

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Bracken, PhD, Study Director — Gynuity Health Projects
Locations (1):
- KEM Hospital, Pune, India

REFERENCES:
- [Derived] Ambardekar S, Shochet T, Bracken H, Coyaji K, Winikoff B. Calibrated delivery drape versus indirect gravimetric technique for the measurement of blood loss after delivery: a randomized trial. BMC Pregnancy Childbirth. 2014 Aug 15;14:276. doi: 10.1186/1471-2393-14-276. PMID 25128176